CLINICAL TRIAL: NCT00799682
Title: An 8 Week, Single Masked, Parallel-Group, Exploratory Study Comparing Ocular Surface Signs and Symptoms in Monotherapy Ocular Hypertension or Glaucoma Patients Randomized to Either Xalatan® or Travatan Z®
Brief Title: Exploratory Study Comparing Signs and Symptoms in Patients With Ocular Hypertension or Glaucoma Using Xalatan R® or Travatan Z®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ophthalmic Consultants of Long Island (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Marguerite McDonald, M.D., Ophthalmic Consultants of Long Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GA6111ZH
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye; Monotherapy for Ocular Hypertension, Glaucoma; Ocular Hypertension; Chronic Open-Angle Glaucoma; Chronic Angle-Closure Glaucoma; Iridotomy; Iridectomy; Pseudo Exfoliate; Pigmentary Glaucoma; Systemic Non-Glaucoma Medications; Hyperemia
MeSH Terms: conditions — Dry Eye Syndromes; Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle; Hyperemia | interventions — Latanoprost; Prostaglandins; Travoprost

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Xalatan® (Active Comparator)
  Interventions: Drug: Xalatan
- Travatan Z® (Active Comparator)
  Interventions: Drug: Travatan Z

INTERVENTIONS:
Drug: Xalatan — 0.005% 1 drop in each eye daily between 7:00 p.m. and 9:00 p.m.
  Other Names: Topical Prostaglandin, Latanoprost Ophthalmic Solution
  Arms: Xalatan®
Drug: Travatan Z — 0.004%, 1 drop in each eye daily between 7:00 p.m. and 9:00 p.m.
  Other Names: Topical Prostaglandin, Travaprost Ophthalmic Solution
  Arms: Travatan Z®

SUMMARY:
The purpose of this study is to determine if there is a difference in the ocular signs and symptoms of subjects' eyes using Xalatan® 0.005% versus Travatan Z® 0.004% based on the outcome of subject assessment and clinical assessment in patients with Ocular Hypertension or Glaucoma with mild to moderate dry eye at baseline in accordance with the Oxford Grading Scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 years of age or older
* Only patients who satisfy all informed consent requirements may be included in the study
* Be likely to complete the entire course of study and comply with study drop regimen, guidelines and visits
* Able to understand drop instructions and instill study drops
* Patients must be on monotherapy for Ocular Hypertension or Glaucoma and agree to a washout period, as according to Appendix E
* Patient has Ocular Hypertension, chronic Open-Angle Glaucoma, chronic Angle-Closure Glaucoma with patent iridotomy/iridectomy, Pseudo Exfoliate Glaucoma, or Pigmentary Glaucoma in each eye at screening visit.
* Patients using systemic non-glaucoma medications known to lower IOP may be included, if on stable dose >30 days prior to screening visit and agree to maintain the regimen throughout the course of the study.
* Patients using non-prescription eye drops or prescription topical eye drops for dry eye may be included, if on stable dose 30 days prior to screening visit and agree to maintain the regimen throughout the course of the study.
* Patients who wear contact lenses with a maintained wearing pattern for the duration of the study
* Best Corrected LogMar VA of ≤0.70 =(20/100 Snellen equivalent)
* Hyperemia Grading ≤2
* IOP ≤ 30 mmHg
* Shirmers 3mm - 9.75mm
* Tear break-up time (TBUT) 4 seconds - 9seconds
* Must meet the Biomicroscopic Criteria for both eyes as defined by the Oxford Grading Scale
* Generally good and stable overall health

Exclusion Criteria:

* Females of childbearing potential (those who are not surgically sterilized or defined as one-year post-menopausal) are excluded from participation in the study if they meet any one of the following conditions:They are currently pregnant,They have a positive result on the urine pregnancy test at the Screening Visit,They intend to become pregnant during the study period,They are breast-feeding,or They are not using highly effective birth control measures:
* Hormonal-oral, implanted, transdermal or injected contraceptives;
* Mechanical-spermicide in conjunction with a barrier such as a condom or diaphragm or IUD Note: All females of childbearing potential must consent to a urine pregnancy test at Screening. Females of childbearing potential are to be instructed to inform the investigator if they become pregnant during the study. Should this occur, the Investigator shall immediately contact the Sponsor. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the patient becomes sexually active during the study, she must agree to use adequate birth control methods as defined above for the remainder of the study.
* Patients who are currently on an investigational agent or discontinued within 30 days prior to the Screening Visit
* Uncontrolled systemic disease
* Patients who have a known medical history of allergy or sensitivity to prostaglandin drugs (topical and/or systemic)
* Patient with any history of refractive surgery
* History of ocular trauma within the past six months in either eye
* History of ocular infection or ocular inflammation within the past three months in either eye
* History of clinically relevant or progressive retinal disease such as retinal degeneration, diabetic retinopathy, or retinal detachment in either eye based on the assessment of the Investigator
* History of any severe ocular pathology according to the Oxford Grading Scale
* greater than Grade 4 dry eye) in either eye
* Intraocular surgery within the past six months as determined by patient history and/or examination in either eye.
* Ocular laser surgery or Punctal Cautery within the past three months as determined by patient history and/or examination in either eye
* Punctal Plugs insertion ≤ 7 days prior to (Visit 1) Screening
* Any abnormality preventing reliable applanation tonometry of either eye.
* Contraindication to pupil dilation or patients with cycloplegia
* Patients with best-corrected visual acuity score worse than 0.70 LogMar (20/100) score in either eye
* Patients with ≤30 days stable dosing regimen before the Screening Visit of any medications or substances administered by any route and used on a chronic basis
* History of Stevens-Johnson Syndrome or Ocular Pemphigoid
* History of liver disease
* Severe clinical vitamin deficiencies or history of vitamin overdose
* Highly variable self-administration of over-the-counter vitamin/herbal products
* Any steroid use within the past 30 days
* Corneal pathology, which could, and of itself, cause an ocular surface disorder
* Visual Field loss which in the opinion of the Investigator is functionally significant or evidence of progress visual field loss within the last year prior to the (Visit 2) Baseline/Randomization
* Patient has a condition or is in a situation which, in the investigator's opinion, may put the subject at a significant risk, may confound study results, or may interfere significantly with the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
OSDI scores (patient's subjective assessment) | Eight Weeks

SECONDARY OUTCOMES:
Clinical Biomicroscopic changes as assessed by Masked Investigator | Eight Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite McDonald, M.D., Principal Investigator — Ophthalmic Consultants of Long Island; Barbara Burger, R.N., Study Director — Ophthalmic Consultans of Long Island
Locations (5):
- United States (5):
  - Ophthalmic Consultants of Long Island, East Meadow, New York
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Ophthalmic Consultants of Long Island, Stony Brook, New York
  - Ophthalmic Consultants of Long Island, Valley Stream, New York